CLINICAL TRIAL: NCT05869188
Title: Effect of Systemic Isotretinoin on Serum Irisin Level in Acne Vulgaris Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Nahed Mohammed Abou Elwfa, Resident, South Valley University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Nahed Abouelwfa
Record Dates: First submitted 2023-05-10; First posted 2023-05-22 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2023-05

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Isotretinoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pateints with Moderate Acne (Active Comparator): 20 patients affected by Acne and More than half of the face is involved. Many papules and pustules, many open or closed comedones. One nodule may be present.
  Interventions: Drug: Isotretinoin
- Pateints with Severe Acne (Active Comparator): 20 patients affected by Acne and Entire face is involved, covered with many papules and pustules, open or closed comedones and rare nodules
  Interventions: Drug: Isotretinoin
- control (Active Comparator): 20 Health participants
  Interventions: Drug: Isotretinoin

INTERVENTIONS:
Drug: Isotretinoin — * Evaluate serum irisin level in acne vulgaris and compare it with healthy control .
  * Evaluate the effect of systemic isotretinoin on serum irisin in acne vulgaris patients .
  Other Names: irisin

SUMMARY:
Acne vulgaris is a chronic inflammatory skin disease affecting the pilosebaceous unit. It is clinically characterized by comedones, papules, pustules, nodules, cysts and scarring on the face and trunk.

The severity of the disease ranges from mild comedonal acne to severe nodulocystic acne which can be permanently disfiguring.In addition to the physical lesions, the disease can have a profound psychologic impact, contributing to low self-esteem, depression and anxiety.In addition to the physical lesions, the disease can have a profound psychologic impact, contributing to low self-esteem, depression and anxiety.

DETAILED DESCRIPTION:
The prevalence of self-reported acne and clinically confirmed acne was 34.69% and 24.39%, respectively. Females reported acne more frequently than males did (39.13% ).The prevalence of clinically confirmed acne was higher among females (28.64%) than males .

Its pathogenesis results from androgen-induced increased sebum production, altered keratinization, inflammation of infundibular epithelium and bacterial colonisation of hair follicles by Propionibacterium acne

There are several treatment modalities for acne vulgaris including topical like topical antibiotics, topical benzoyl peroxide, topical azelaic acid and topical retinoids. Systemic therapy like antibiotics, hormonal therapy and isotretinoin .

Adipokines may have a role in the pathogenesis of acne vulgaris and are associated with acne severity. Irisin, a hormone -like myokine, is one of the adipokines with anti- inflammatory and anti-oxidant effects

There is limited evidence for physical modalities (e.g., laser therapy, light therapy, chemical peels) and complementary therapies (e.g., purified bee venom, low-glycemic-load diet, tea tree oil) .

isotretinoin (13-cis retinoic acid) is the most potent known inhibitor of sebum production. The multiple modes of action for isotretinoin includs suppression of sebaceous gland activity, normalization of the pattern of keratinization within the sebaceous gland follicle, inhibition of inflammation and reduction of growth of Propionibacterium acne .

ELIGIBILITY:
Inclusion Criteria:

* Cases with moderate and severe acne.
* Clinical diagnosis of acne Disease
* Patient not receive any treatment for acne vulgaris at least six months duration.

Exclusion Criteria:

1 Pregnant and lactating women. 2. History of chronic liver disease . 3. Cardiovascular disorders . 4. Renal disease . 5. Hyperlipidemia . 6. Depression or mental illness. 7. Insulin dependent diabetes 8 Thyroid disease. 9 Osteoporosis or low bone mineral density . 10 Intestinal disorders such as inflammatory bowel disease or ulcerative colitis

Ages: 14 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Evalaute serum level of irisin in acne patient | From 0 base to 3 Months from starting the treatment Day
  Assessment of clinical improvement according to:(8) G4(excellent:100% reduction) G3(good:75-99% reduction) G2(moderate: 50-74% reduction) G1(insufficient :1-49% reduction) G0(unchanged) G-1(worse)

SECONDARY OUTCOMES:
Evalaute the effect of treatment with systemic isotretinon | From 0 base to 3 Months from starting the treatment Day
  Evalaute the effect of treatment with systemic isotretinon on the level of serum irisin .

CONTACTS AND LOCATIONS:
Overall Officials: Essra Abass, Lecturer, Principal Investigator — Clinical Pathology Department, Faculty of Medicine, South valley University
Locations (1):
- Qena Hospital, Qina, Egypt